CLINICAL TRIAL: NCT00436072
Title: Phase I Study of ZD6474, Cetuximab, and Irinotecan in Patients With Metastatic Colorectal Cancer
Brief Title: ZD6474, Cetuximab, and Irinotecan in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Jeffrey A. Meyerhardt, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-177
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Cancer
Keywords: ZD6474; cetuximab; irinotecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — vandetanib; Cetuximab; Irinotecan

INTERVENTIONS:
Drug: ZD6474 — Orally on a daily basis
Drug: Cetuximab — Infusion once weekly
Drug: Irinotecan — Infusion once the safe dose of ZD6474 and cetuximab is established

SUMMARY:
This research study will test the safety of the investigational drug, ZD6474, in combination with 2 other drugs that are standard in the treatment of colon and rectal cancer (cetuximab and irinotecan). ZD6474 blocks the action of two substances in the body: vascular endothelial growth factor receptor (VEGFR) and epidermal growth factor receptor (EGFR). VEGFR stimulates the formation of new blood vessels. When cancer cells produce VEGFR, new blood vessels are made that provide blood to the cancer cells. The blood carries nutrients and oxygen, allowing the cancer cells to live and grow. EGFR controls how quickly cells grow and multiply. Both of these substances are found on normal cells, but they are found in much higher levels on cancer cells.

DETAILED DESCRIPTION:
* The main purpose is to find the highest dose of ZD6474 that is safe to give in combination with cetuximab and irinotecan. We will also be collecting information on how the body responds to the study drugs and what effects, good or bad, it has on treatment of colon and rectal cancer.
* Initially we plan to add ZD6474 to cetuximab alone. Small groups of participants will be enrolled in steps. The first group will be given a certain dose of ZD6474 and cetuximab. If the participants have few or manageable side effects, the next small group of people will receive a higher dose of ZD6474. This increase will continue until the study doctors find the highest dose that can be given.
* Once we determine the highest dose of ZD6474 with cetuximab, we will add irinotecan at increasing doses to determine the safety of all three drugs combined. The participant will know whether they are receiving the two or three drug combination.
* In order to confirm the safety of combining these drugs and to understand more how they work and interact with each other, some participants on this study will take just the ZD6474 for 2 weeks prior to starting the cetuximab and/or irinotecan.
* Each cycle of treatment is 8 weeks long. All participants will start taking ZD6474 orally, on day one and continue taking it at home thereafter. Cetuximab and irinotecan are given intravenously. Cetuximab is given once a week. Irinotecan will be given to participants that enter the trial once the safe dose of ZD6474 and cetuximab is determined. Irinotecan is given on Day 15 of cycle one, then every other week.
* Participants will be asked to visit the clinic every week for the first three weeks they are on the study. After the first three weeks, they will be required to visit with the doctor every other week. These visits will include physical exams, routine blood tests, scans, and other tests or procedures to monitor health.
* In addition to routine blood tests, blood tests for research will be done on the last 10 subjects on the trial. Test results from this sample will be used to evaluate the participants condition.
* In order to be treated on this study, a tumor tissue specimen must ba available for research testing. The specimen will be taken from a biopsy that was done before the participant enrolled on the study.
* Participants can continue on the study drug as long as they tolerate the drug and the cancer does not grow.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic colorectal cancer
* 1-2 prior therapies for metastatic colorectal cancer. Prior adjuvant therapy not included in the number of priors unless recurrence within 12 months of last dose of therapy and then the adjuvant therapy will be counted.
* Tumor is K-ras wildtype by method of choice at respective institution (testing codons 12 and 13)
* Measurable disease according to the RECIST criteria
* 18 years of age or older
* ECOG Performance Status of 0-2
* Completed any major surgery 4 weeks from registration and any minor surgery 2 weeks from registration
* Adequate bone marrow function
* Adequate renal function
* Adequate hepatic function
* Normal range of serum calcium and magnesium
* Agree to use an effective form of contraception during the study and 90 days following the last dose of medication
* Negative urine or serum pregnancy test

Exclusion Criteria:

* History of prior malignancy within the past 3 years except curatively treated basal cell carcinoma of the skin, cervical intra-epithelial neoplasia, or treated localized prostate cancer
* Prior therapy with gefitinib, erlotinib, cetuximab, ABX-EGF or other specific EGFR inhibitor
* Known hypersensitivity to any components of each drug
* Pregnant or lactating women
* Any other medical condition, including mental illness or substance abuse, deemed by the clinician to be likely to interfere
* Potassium < 4.0 mEg/L despite supplementation
* Evidence of severe or uncontrolled systemic disease or any concurrent illness that, in the opinion of the investigator, makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Clinically significant cardiac event such as myocardial infarction: NYHA classification of heart disease greater than or equal to 2 that, in the opinion of the investigator, increases the risk of ventricular arrhythmia within 3 months before entry; or presence of cardiac disease
* History of arrythmia which is symptomatic or requires treatment or asymptomatic sustained ventricular tachycardia
* Previous history of QTc prolongation as a result from other medication that required discontinuation of that medication
* Congenital long QT syndrome, or 1st degree relative with unexplained sudden death under 40 years of age
* Presence of left bundle branch block
* QTc with Bazett's correction that is unmeasurable , or greater then 480msec on screening ECG
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function
* Hypertension not controlled by medical therapy
* Patients lacking physical integrity of the upper gastrointestinal tract or who have malabsorption syndrome
* Currently active diarrhea that may affect patient's ability to absorb ZD6474 or tolerate potential diarrhea from study drugs
* For patients entering dose levels 4-6, prior history of irinotecan toxicity requiring a dose reduction lower than the dose of irinotecan that the patient will be receiving on this study
* Receipt of any investigational agents within 30 days prior to commencing study treatment
* Last dose of prior chemotherapy or radiation therapy discontinued less thn 4 weeks before the start of study therapy
* Incompletely healed surgical incisions, at the discretion of the investigator
* Any unresolved toxicity greater than CTC grade 1 from previous anti-cancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2007-02; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To determine the tolerability and maximum tolerated dose of combining ZD6474, cetuximab and irinotecan in patients with metastatic colorectal cancer refractory to prior cytotoxic chemotherapy. | Years

SECONDARY OUTCOMES:
Determine response rate, progression-free survival and overall survival of adding ZD6474 to cetuximab and irinotecan in this patient population. | Years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Meyerhardt, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

REFERENCES:
- [Result] Meyerhardt JA, Ancukiewicz M, Abrams TA, Schrag D, Enzinger PC, Chan JA, Kulke MH, Wolpin BM, Goldstein M, Blaszkowsky L, Zhu AX, Elliott M, Regan E, Jain RK, Duda DG. Phase I study of cetuximab, irinotecan, and vandetanib (ZD6474) as therapy for patients with previously treated metastastic colorectal cancer. PLoS One. 2012;7(6):e38231. doi: 10.1371/journal.pone.0038231. Epub 2012 Jun 12. PMID 22701615